CLINICAL TRIAL: NCT05628714
Title: Effectiveness of a Patient Decision Aid for Patients With Superficial Basal Cell Carcinoma: a Pre- and Post-implementation Study
Brief Title: A Patient Decision Aid for Patients With Superficial Basal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Catharina Ziekenhuis Eindhoven (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-0624
Record Dates: First submitted 2022-11-08; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Superficial Basal Cell Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Patients who did not use the PDA
- PDA-group: Patients who did use the PDA
  Interventions: Other: Patient decision aid for patients with superficial basal cell carcinoma

INTERVENTIONS:
Other: Patient decision aid for patients with superficial basal cell carcinoma — An online WebApp
  Other Names: PDA
  Groups: PDA-group

SUMMARY:
A patient decision aid (PDA) was tested in a population of patients with superficial basal cell carcinoma. This study evaluates whether the use of a PDA improved outcomes like decisional conflict and knowledge.

DETAILED DESCRIPTION:
Background Patients with a superficial basal cell carcinoma (sBCC) can choose between several treatment options with specific advantages and disadvantages. A patient decision aid (PDA) might facilitate a personalized decision.

Objectives This study evaluates whether the use of a PDA results in a decreased level of decisional conflict, improved satisfaction with the treatment decision, and increased knowledge on prevention, recognition of BCC, and treatment options.

Methods A prospective multicentre pre- and post-implementation study was performed amongst patients with a newly diagnosed sBCC comparing a group that did not use the PDA (control group) with a group that did (PDA group). The primary outcome was the level of decisional conflict measured by the total mean score on the 'decisional conflict scale' (DCS) directly before treatment. Higher scores correspond with higher levels of decisional conflict (scale 0-100). Knowledge of disease and treatment options was evaluated by using a questionnaire.

Results Questionnaires were completed by 103 patients in the control group and 109 patients in the PDA group. The mean total score on the DCS in the control group was 22.78 (SD 14.76) compared to 22.34 (SD 14.54) in the PDA group. The adjusted mean difference was -0.39 (95% CI -4.47-3.70, p=0.851). Cohen's effect size for the total score on the DCS was 0.03. Use of the PDA resulted in a significant increase of knowledge on recognition of BCC (p<0.001) and treatment options for sBCC (p=0.005). According to exploratory subgroup analyses the unadjusted mean difference in DCS score was higher in patients with sBCC in the head and neck area (-4.53, p=0.378), patients without a history of BCC (-3.76, p=0.251), and patients with higher educational level (-4.71, p=0.196).

Conclusion In the total study population with newly diagnosed sBCC, use of a PDA increased knowledge on relevant issues, but had no significant effect on the level of decisional conflict when compared with a control group. Exploratory subgroup analyses suggest that specific subgroups of patients may benefit from the use of a PDA, but these results need to be verified in larger studies.

ELIGIBILITY:
Inclusion criteria:

* patients older than 18 years
* patients with a clinically or histologically confirmed sBCC

Exclusion criteria:

- patients that could not read (Dutch)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * patients older than 18 years
  * patients that could read (Dutch)
  * patients with a clinically or histologically confirmed sBCC
Sampling Method: Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Decisional conflict | Before treatment
  The primary outcome was the level of decisional conflict measured by the total mean score on the 'decisional conflict scale' (DCS) directly before treatment. Higher scores correspond with higher levels of decisional conflict (scale 0-100).

SECONDARY OUTCOMES:
Knowledge | Before treatment
  To evaluate patient knowledge, we used a questionnaire adapted by our research group from a knowledge assessment for melanoma. [14, 15] (Appendix B) The questionnaire included items on sun-protection (7 statements), risk factors for developing a BCC (10 statements), treatment options for sBCC (7 statements), and ways to recognize a BCC (6 statements). The proportions of patients with correct answers (true/false) for all statements within a domain were compared between the two groups.
Patient satisfaction | 3 Months post-treatment
  Patient satisfaction with treatment decision was measured using the mean scores on the subscale 'effective decision making' and separate questions of this subscale of the DCS at 3 months post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No